CLINICAL TRIAL: NCT05472363
Title: Electroencephalogram Coupled Non-invasive Brain Stimulation For Assessment of Cortical Excitability
Brief Title: TMS-EEG for Cortical Excitability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges in TMS-EEG data protocol optimization
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zafer Keser, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-012185
Record Dates: First submitted 2022-07-07; First posted 2022-07-25 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Acquired Brain Injury; Stroke; Traumatic Brain Injury; Healthy
MeSH Terms: conditions — Brain Injuries; Stroke; Brain Injuries, Traumatic | interventions — Electroencephalography; Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non-Stroke Subjects (Experimental): Subjects will receive up to 30 minutes of focal simulation with either TMS or tDCS administered to one brain location within standard safety protocols
  Interventions: Diagnostic Test: Electroencephalogram; Procedure: Transcranial Magnetic Stimulation; Procedure: Transcranial Direct Current Stimulation
- Stroke Subjects (Experimental): Subjects will receive up to 30 minutes of focal stimulation with either TMS or tDCS administered to one brain location within standard safety protocols
  Interventions: Diagnostic Test: Electroencephalogram; Procedure: Transcranial Magnetic Stimulation; Procedure: Transcranial Direct Current Stimulation

INTERVENTIONS:
Diagnostic Test: Electroencephalogram — A routine test that involves attaching small wires to the head to read the electrical activity of the brain
  Other Names: EEG
Procedure: Transcranial Magnetic Stimulation — Noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain. An electromagnetic coil is placed against the scalp near the forehead. The electromagnet painlessly delivers repetitive magnetic pulses to simulate nerve cells in the brain.
  Other Names: TMS
Procedure: Transcranial Direct Current Stimulation — Noninvasive procedure that uses direct electrical currents to stimulate the brain. A constant, low intensity current is passed through two electrodes that are place on the head.
  Other Names: tDCS

SUMMARY:
This research study is being done to look at the safety and diagnostic benefit of conducting an TMS(transcranial magnetic stimulation)-EEG measured before and after a brief experimental stimulation session using investigational devices repetitive TMS or transcranial direct current stimulation (tDCS).

ELIGIBILITY:
Inclusion Criteria - Stroke:

- Acquired brain injury such as ischemic or hemorrhagic stroke or traumatic brain injury.

Inclusion Criteria - Healthy Controls:

- No known active neurological disorder.

Exclusion Criteria - Stroke:

* Pregnancy
* Contraindication to MRI or TMS including metallic implanted objects.
* Medical instability or inability to cooperate during the study as assessed by the treating physician to participate in the study.
* Severe aphasia.
* History of epilepsy.
* History of active depression or treatment resistant depression.
* History of schizophrenia.

Exclusion Criteria - Healthy Controls:

* Pregnancy
* Contraindication to MRI or TMS including metallic implanted objects.
* History of acquired brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Western Aphasia Battery (WAB) Aphasia (AQ) and Language Quotients (LQ) | Baseline, 3 months
  Measured using Western Aphasia Battery Bedside Version. Higher score is better. Ranged from 0-100.
Change in Modified Rankin Scale | Baseline, 3 months
  Measured using the Modified Rankin Scale (MRS) to assess functional outcome measure in stroke that utilizes a structured interview to assign subjects MRS grades 0-5 in a systematic way, grade 5 is severe disability, grade 0 is no symptoms at all
Change in neurological outcome (NIHSS) | Baseline, 3 months
  Measured using the National Institutes of Health Stroke Scale (NIHSS). 15-item test to assess stroke-related neurologic deficits, each item scored with 3-5 grades with 0 as normal.
EEG and TMS-EEG functional connectivity | Baseline
  EEG power in high and low frequency bands will be measured and power density maps will be created. TMS-evoked potentials and oscillations will be measured.
MRI based structural connectivity. | Baseline
  Microstructural integrity of the networks will be quantified by using diffusion weighted imaging metrics such as mean diffusivity.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Keser, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials